CLINICAL TRIAL: NCT03230695
Title: Effects of Robotic Therapy and Transcranial Direct Current Stimulation on Motor Performance of the Paretic Upper Limb in the Early Phase After Stroke
Brief Title: Robotic Therapy and Brain Stimulation in the Early Phase After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RCT2129001
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Stroke
Keywords: stroke; robotic therapy; transcranial direct current stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation + robotic therapy (Active Comparator): Active transcranial direct current stimulation will be applied during 20 minutes prior to robotic training.
  Number of interventions sessions: 1
  Interventions: Device: Robotic Therapy; Device: Active stimulation
- Sham stimulation + robotic therapy (Sham Comparator): Sham transcranial direct current stimulation will be applied during 20 minutes prior to robotic training.
  Number of interventions sessions: 1
  Interventions: Device: Robotic Therapy; Device: Sham stimulation

INTERVENTIONS:
Device: Robotic Therapy — Robotic therapy (MIT - Manus, Interactive Motion Technologies) will be administered for 40 minutes to the paretic upper limb.
Device: Active stimulation — Active transcranial direct current stimulation will be applied with the cathode positioned over the ipsilesional primary motor cortex and the anode over the contralateral supraorbital region for 20 minutes (1mA).
  Arms: Active stimulation + robotic therapy
Device: Sham stimulation — In sham transcranial direct current stimulation, no current will be delivered through the transcranial direct current stimulation device after the first 30 seconds.
  Arms: Sham stimulation + robotic therapy

SUMMARY:
Stroke is the second cause of death worldwide and the majority of the survivors remain with motor impairments. Inhibition of the motor cortex of the unaffected hemisphere has emerged as a potential intervention to enhance effects of other rehabilitation strategies on improvement of motor performance of the paretic upper limb. In this proof-of-concept study we will evaluate the effects of inhibition of the motor cortex of the unaffected hemisphere associated with robotic therapy on improvement of motor performance of the paretic upper limb in the early phase post-stroke.

DETAILED DESCRIPTION:
The main goal of this study is to test the proof of concept of benefits of inhibition of the motor cortex of the unaffected hemisphere on learning evaluated by improvement in kinematics of motor performance, in patients with upper limb paresis in the early phase post-stroke. For this purpose, patients will be randomized to receive real or sham transcranial direct current stimulation before a session of robotic therapy. Data will be collected by kinematic assessment performed automatically by the robot at baseline, immediately after and 24h after the intervention.

The working hypothesis is that one session of upper limb motor training will lead to improvement of performance in metrics of kinematics, and this improvement will be maintained up to 24h after the end of the training.

ELIGIBILITY:
Inclusion Criteria:

Ischemic or hemorrhagic stroke onset from 3 days to 9 weeks before, confirmed by computed tomography or magnetic resonance imaging.

Motor impairment of an upper limb, defined as a score between 1 - 3 in the Medical Research Council Scale, for at lest one the following movements: elbow extension, shoulder flexion, or shoulder extension.

Ability to provide written informed consent.

Ability to comply with the schedule of interventions and evaluations in the protocol.

Exclusion Criteria:

Severe spasticity at the paretic elbow, wrist or fingers, defined as a score of > 3 in the Modified Ashworth Spasticity Scale.

No active shoulder and elbow movements

Uncontrolled medical problems such as end-stage cancer or renal disease

Pregnancy

Potential contraindications to transcranial direct current stimulation: history of seizures, lesions on the scalp, intracranial metal implants, prior intracranial surgery, use of drugs that interfere on cortical excitability (such as antiepileptic drugs, benzodiazepines)

Other neurological disorders such as Parkinson's disease

Psychiatric illness

Aphasia or severe cognitive deficits that compromise comprehension of the experimental protocol or ability to provide consent.

Hemineglect

Cerebellar lesions or on cerebellar pathways

Contact precautions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-08-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Movement Smoothness | Kinematic assessment at baseline, immediately after intervention; and 24h after.
  The speed shape, calculated as mean speed divided by peak speed.

SECONDARY OUTCOMES:
Number of peaks of the movement | kinematic assessment at baseline, immediately after intervention; and 24h after.
  Number of peaks of the movement is calculated as the negative of the number of peaks in the speed profile.
Jerk metric of the movement | kinematic assessment at baseline, immediately after intervention; and 24h after
  Jerk metric of the movement is calculated by dividing the negative mean jerk magnitude by the peak speed.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana B Conforto, D, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Suzana Bleckmann Reis, São Paulo, Brazil